CLINICAL TRIAL: NCT06189248
Title: The Effects of Resourcefulness Intervention Group on the Interpersonal Competence, Relationship Adjustment, and Negative Emotion in College Students.
Brief Title: The Effects of Resourcefulness Intervention Group
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chien Yu Lai, Clinical Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022RI
Record Dates: First submitted 2023-08-04; First posted 2024-01-03 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Health Resources

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 6 group activities designed with resourcefulness skills will be performed in the intervention group.
  1. Introduction of Resourcefulness
  2. Issue of the Interpersonal Competence: Applications of both personal and social resourcefulness strategies
  3. Issues of the Interpersonal Competence & Relationship Adjustment: Applications of both personal and social resourcefulness strategies
  4. Issue of the Relationship Adjustment: Applications of both personal and social resourcefulness strategies
  5. Issue of the Negative Emotion: Applications of both personal and social resourcefulness strategies
  6. Conclusion
  Interventions: Behavioral: Resourcefulness intervention
- Observation group (No Intervention): No intervention for the observation group.

INTERVENTIONS:
Behavioral: Resourcefulness intervention — Teaching personal and social resourcefulness skills.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to analyze the effects of resourcefulness interventions on interpersonal competence, relationship adjustment, and negative emotion in young adults. An interventional and longitudinal study design will be used to design resourcefulness intervention groups and examine the effects of resourcefulness group interventions on interpersonal competence, relationship adjustment, and negative emotion in young adults.

DETAILED DESCRIPTION:
Purposes: To analyze the effects of resourcefulness interventions on interpersonal competence, relationship adjustment, and negative emotion in young adults.

Methods: The interventional and longitudinal study design will be used in this study. The resourcefulness intervention groups will be built up and the effects of resourcefulness group interventions on interpersonal competence, relationship adjustment, and negative emotion in young adults will be examined.

Anticipated results: the study results will be important references for interpersonal and intimate relationship counseling for college students.

ELIGIBILITY:
Inclusion Criteria:

Participants who have ever had at least one experience in the relationship.

Exclusion Criteria:

1. The ones who are taking continuous education in the evening.
2. The ones who have been diagnosed with major depressive disorder, panic disorder, or other psychotic diseases which influenced cognitive functions.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Resourcefulness Scale | Four times, T0 pretest, T1 six weeks later, T2 three months later, T3 six months. From date of first documented progression, assessed up to 7.5 months.
  The levels of resourcefulness
Interpersonal Competence Questionnaire | Four times, T0 pretest, T1 six weeks later, T2 three months later, T3 six months. From date of first documented progression, assessed up to 7.5 months.
  The levels of interpersonal competence
Relationship Adjustment Scale | Four times, T0 pretest, T1 six weeks later, T2 three months later, T3 six months. From date of first documented progression, assessed up to 7.5 months.
  The adjustment situation in the relationship
State-Trait Anxiety Inventory-S | Four times, T0 pretest, T1 six weeks later, T2 three months later, T3 six months. From date of first documented progression, assessed up to 7.5 months.
  The levels of anxiety
Center for Epidemiological Studies National Institute of Mental Health-Depression Scales | Four times, T0 pretest, T1 six weeks later, T2 three months later, T3 six months. From date of first documented progression, assessed up to 7.5 months.
  The levels of depression

CONTACTS AND LOCATIONS:
Overall Officials: Chien Yu Lai, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- NTUNHS, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No